CLINICAL TRIAL: NCT05065983
Title: A Phase 2 Open-Label Study to Assess the Safety and Immunogenicity of PXVX0317 (Chikungunya Virus Virus-Like Particle Vaccine [CHIKV VLP], Aluminum Hydroxide Adjuvanted)
Brief Title: A Study to Assess the Safety and Immunogenicity of PXVX0317 Chikungunya Virus Virus-Like Particle Vaccine
Acronym: CHIKV VLP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EBSI-CV-317-010
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Chikungunya Virus

STUDY DESIGN:
Intervention Model Description: Open Label Safety and Immunogenicity
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PXVX0317 (CHIKV VLP, alum-adjuvanted) vaccine (Experimental): All study participants will receive the same Investigational Product (40 µg CHIKV VLP, alum-adjuvanted according to the same single dose schedule on Day 1).
  Interventions: Biological: CHIKV VLP, adjuvanted

INTERVENTIONS:
Biological: CHIKV VLP, adjuvanted — Adjuvanted formulation includes aluminum hydroxide

SUMMARY:
The objective of this study is to assess the safety and immunogenicity of PXVX0317 (Chikungunya Virus Virus-Like Particle Vaccine [CHIKV VLP], aluminum hydroxide adjuvanted).

DETAILED DESCRIPTION:
Primary Objectives:

1. To assess the induction of anti-CHIKV neutralizing antibody responses following a single adjuvanted dose of PXVX0317 (40 µg CHIKV VLP, alum-adjuvanted) as measured 21 days (Day 22) after vaccination.
2. To assess the induction of anti-CHIKV neutralizing antibody responses following a single adjuvanted dose of PXVX0317 as measured 7 days (Day 8), 14 days (Day 15), and 56 days (Day 57) after vaccination.

Secondary Objectives:

1. To assess safety of a single adjuvanted dose of PXVX0317 in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent voluntarily signed by participant.
2. Any gender, 18 to 45 years of age (inclusive).
3. Generally healthy, in the opinion of the Investigator, based on medical history, physical examination, and screening laboratory assessments.
4. Women who are either:

   (i). Not of childbearing potential (CBP): pre-menarche, anatomically sterile, or post-menopausal (defined as ≥12 months without menses) or (ii). Meeting all the following criteria: Negative urine pregnancy test at screening visit; and Negative urine pregnancy test immediately prior to dosing at Day 1; and using an acceptable method of contraception (if female of childbearing potential) for the duration of participation, such as: Hormonal contraceptives (e.g., implants, pills, patches) initiated ≥ 30 days prior to dosing or; Intrauterine device (IUD) inserted ≥30 days prior to dosing or; double barrier type of birth control (male condom with female diaphragm, male condom with cervical cap).

Exclusion Criteria:

1. Currently pregnant, breastfeeding, or planning to become pregnant during the study.
2. Body Mass Index (BMI) ≥35 kg/m2.
3. Positive laboratory evidence of current infection with human immunodeficiency virus (HIV-1, HIV-2), hepatitis C virus (HCV) or hepatitis B virus (HBV).
4. History of severe allergic reaction or anaphylaxis to any component of the investigational product (IP).
5. History of known congenital or acquired immunodeficiency that could impact response to vaccination (e.g., leukemia, lymphoma, generalized malignancy, functional or anatomic asplenia, alcoholic cirrhosis).
6. Prior or anticipated receipt of immunomodulatory or immunosuppressive therapy from six months prior to screening through Day 64.
7. Receipt or anticipated receipt of blood or blood-derived products from 90 days prior to screening through Day 64.
8. Acute disease within the last 14 days (participants with an acute mild febrile illness can be considered for a deferral of vaccination two weeks after the illness has resolved and treatment has been completed).
9. Clinically significant cardiac, pulmonary, respiratory, rheumatologic, or other chronic disease, in the opinion of the Investigator. This may include chronic illness requiring hospitalization in the last one month prior to screening.
10. Enrollment in an interventional study and/or receipt of another investigational product from 30 days prior to screening through the duration of study participation.
11. Receipt or anticipated receipt of any vaccine from 30 days prior to screening through Day 64.
12. Prior receipt of an investigational CHIKV vaccine/product.
13. Detectable baseline anti-CHIKV IgG antibody as determined by ELISA.
14. Any other condition that, in the opinion of the investigator, could adversely impact the participant's participation or the conduct of the study, creates an unacceptable risk to the participant, or may interfere with the conduct of the study or validity of the data.
15. Restricted venous access that would prevent the collection of plasma and serum necessary for participation.
16. Weight <110 pounds.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ajiboye, Study Director — Emergent BioSolutions
Locations (1):
- Johnson County ClinTrials, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 1 U.S. site.
Period: Overall Study
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Started | 25
Exposed (Screened participants who received study vaccination.) | 25
Safety (Participants who received study vaccination and provided safety assessment data.) | 25
mITT (Modified Intent-to-treat Population = All participants who were vaccinated and had at least one post injection anti-CHIKV SNA NT80 result.) | 25
Completed | 23
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Day 1 predose (baseline) geometric mean anti-chikungunya luciferase neutralizing antibody titer. [Geometric Mean (Full Range); unit: Titer] — Day 1 predose (baseline) geometric mean anti-chikungunya luciferase neutralizing antibody titer. Values below the lower limit of quantitation of 15 were imputed as half the lower limit of quantitation or 7.5.
  Titer | 7.5 [7.5 to 7.5]

OUTCOME MEASURES:

1. Primary Outcome: CHIKV SNA (Serum Neutralizing Antibody) Seroresponse Rate at Day 22
Description: CHIKV SNA Seroresponse Rate (Titer >=40) and Associated 95% Confidence Interval (CI) at Day 22
Time Frame: 21 days post vaccination
Population: mITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Percentage of participants | 100.0 [86.7 to 100.0]

2. Primary Outcome: CHIKV SNA GMT (Geometric Mean Titer) at Day 22
Description: CHIKV SNA GMT and Associated 95% CI at Day 22
Time Frame: 21 days post vaccination
Population: mITT
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Titer | 2365.2 [1625.0 to 3442.4]

3. Primary Outcome: CHIKV SNA Seroresponse Rates at Days 8, 15, and 57
Description: CHIKV SNA Seroresponse Rates with Associated 95% CIs at Days 8, 15, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Percentage of participants
  Day 8 titer at or above 40 | 76.0 [56.6 to 88.5]
  Day 15 titer at or above 40 | 100.0 [86.7 to 100.0]
  Day 57 titer at or above 40: number analyzed (Participants) | 24
  Day 57 titer at or above 40 | 100.0 [86.2 to 100.0]

4. Primary Outcome: CHIKV SNA GMTs at Days 8, 15, and 57
Description: CHIKV SNA GMTs with Associated 95% CIs at Days 8, 15, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Titer
  Day 8 | 117.4 [68.3 to 201.8]
  Day 15 | 1397.1 [901.9 to 2164.2]
  Day 57: number analyzed (Participants) | 24
  Day 57 | 1069.7 [720.2 to 1588.9]

5. Primary Outcome: CHIKV ELISA (Enzyme-Linked Immunosorbent Assay) IgG GMTs at Days 8, 15, 22, and 57
Description: CHIKV ELISA IgG GMTs with Associated 95% CIs at Days 8, 15, 22, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Titer
  Day 8 | 0.71 [0.66 to 0.77]
  Day 15 | 1.1 [0.88 to 1.4]
  Day 22 | 1.5 [1.3 to 1.9]
  Day 57: number analyzed (Participants) | 24
  Day 57 | 1.2 [1.0 to 1.4]

6. Primary Outcome: CHIKV ELISA IgM GMTs at Days 8, 15, 22, and 57
Description: CHIKV ELISA IgM GMTs with Associated 95% CIs at Days 8, 15, 22, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Titer
  Day 8 | 1.2 [0.93 to 1.6]
  Day 15 | 5.0 [4.0 to 6.3]
  Day 22 | 6.2 [5.0 to 7.7]
  Day 57: number analyzed (Participants) | 24
  Day 57 | 2.9 [2.1 to 3.8]

7. Primary Outcome: Geometric Mean Fold Increase (GMFI) in CHIK SNA Titers at Days 8, 15, 22, and 57
Description: GMFI in CHIK SNA Titers from Day 1 to Days 8, 15, 22, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Fold increase
  Day 8 | 15.6 [9.1 to 26.9]
  Day 15 | 186.3 [120.3 to 288.6]
  Day 22 | 315.4 [216.7 to 459.0]
  Day 57: number analyzed (Participants) | 24
  Day 57 | 142.6 [96.0 to 211.9]

8. Primary Outcome: GMFI in CHIK ELISA IgG at Days 8, 15, 22, and 57
Description: GMFI in CHIK ELISA IgG from Day 1 to Days 8, 15, 22, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Fold increase
  Day 8 | 0.93 [0.77 to 1.1]
  Day 15 | 1.4 [1.0 to 2.0]
  Day 22 | 2.0 [1.5 to 2.6]
  Day 57: number analyzed (Participants) | 24
  Day 57 | 1.7 [1.4 to 2.1]

9. Primary Outcome: GMFI in CHIK ELISA IgM at Days 8, 15, 22, and 57
Description: GMFI in CHIK ELISA IgM from Day 1 to Days 8, 15, 22, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Fold increase
  Day 8 | 3.1 [2.3 to 4.1]
  Day 15 | 12.6 [9.9 to 16.1]
  Day 22 | 15.6 [12.6 to 19.4]
  Day 57: number analyzed (Participants) | 24
  Day 57 | 7.2 [5.3 to 9.8]

10. Primary Outcome: Number and Percentage of Participants With a CHIKV SNA Titer at or Above Threshold Values at Days 8, 15, 22, and 57
Description: Number and Percentage of Participants with a CHIKV SNA Titer ≥15, 40, 60, 80, 100, 160, 640, and 4-fold Rise Over Baseline Thresholds at Days 8, 15, 22, and 57
Time Frame: 56 days post vaccination
Population: mITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Percentage of participants
  Day 8 : Titer at or above 15 | 96.0 [80.5 to 99.3]
  Day 8 : Titer at or above 40 | 76.0 [56.6 to 88.5]
  Day 8 : Titer at or above 60 | 68.0 [48.4 to 82.8]
  Day 8 : Titer at or above 80 | 56.0 [37.1 to 73.3]
  Day 8 : Titer at or above 100 | 52.0 [33.5 to 70.0]
  Day 8 : Titer at or above 160 | 48.0 [30.0 to 66.5]
  Day 8 : Titer at or above 640 | 12.0 [4.2 to 30.0]
  Day 8 : Titer at or above 4-fold rise over baseline | 88.0 [70.0 to 95.8]
  Day 15 : Titer at or above 15 | 100.0 [86.7 to 100.0]
  Day 15 : Titer at or above 40 | 100.0 [86.7 to 100.0]
  Day 15 : Titer at or above 60 | 100.0 [86.7 to 100.0]
  Day 15 : Titer at or above 80 | 100.0 [86.7 to 100.0]
  Day 15 : Titer at or above 100 | 100.0 [86.7 to 100.0]
  Day 15 : Titer at or above 160 | 96.0 [80.5 to 99.3]
  Day 15 : Titer at or above 640 | 76.0 [56.6 to 88.5]
  Day 15 : Titer at or above 4-fold rise over baseline | 100.0 [86.7 to 100.0]
  Day 22 : Titer at or above 15 | 100.0 [86.7 to 100.0]
  Day 22 : Titer at or above 40 | 100.0 [86.7 to 100.0]
  Day 22 : Titer at or above 60 | 100.0 [86.7 to 100.0]
  Day 22 : Titer at or above 80 | 100.0 [86.7 to 100.0]
  Day 22 : Titer at or above 100 | 100.0 [86.7 to 100.0]
  Day 22 : Titer at or above 160 | 96.0 [80.5 to 99.3]
  Day 22 : Titer at or above 640 | 92.0 [75.0 to 97.8]
  Day 22 : Titer at or above 4-fold rise over baseline | 100.0 [86.7 to 100.0]
  Day 57 : Titer at or above 15: number analyzed (Participants) | 24
  Day 57 : Titer at or above 15 | 100.0 [86.2 to 100.0]
  Day 57 : Titer at or above 40: number analyzed (Participants) | 24
  Day 57 : Titer at or above 40 | 100.0 [86.2 to 100.0]
  Day 57 : Titer at or above 60: number analyzed (Participants) | 24
  Day 57 : Titer at or above 60 | 100.0 [86.2 to 100.0]
  Day 57 : Titer at or above 80: number analyzed (Participants) | 24
  Day 57 : Titer at or above 80 | 100.0 [86.2 to 100.0]
  Day 57 : Titer at or above 100: number analyzed (Participants) | 24
  Day 57 : Titer at or above 100 | 100.0 [86.2 to 100.0]
  Day 57 : Titer at or above 160: number analyzed (Participants) | 24
  Day 57 : Titer at or above 160 | 95.8 [79.8 to 99.3]
  Day 57 : Titer at or above 640: number analyzed (Participants) | 24
  Day 57 : Titer at or above 640 | 75.0 [55.1 to 88.0]
  Day 57 : Titer at or above 4-fold rise over baseline: number analyzed (Participants) | 24
  Day 57 : Titer at or above 4-fold rise over baseline | 100.0 [86.2 to 100.0]

11. Secondary Outcome: Incidence of Solicited Adverse Events (AE) Through Day 8
Description: Incidence of Solicited AEs Through Day 8
Time Frame: 7 days post vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Participants
  Any solicited AE | 17
  Any systemic solicited AE | 12
  Fever | 1
  Chills | 1
  Fatigue | 8
  Headache | 7
  Myalgia | 5
  Arthralgia | 2
  Nausea | 2
  Any local solicited AE | 14
  Injection site pain | 14
  Injection site redness | 0
  Injection site swelling | 0

12. Secondary Outcome: Incidence of Unsolicited AEs Through Day 29
Description: Incidence of Unsolicited AEs Through Day 29
Time Frame: 28 days post vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Participants
  Participants with any unsolicited AEs | 8
  General disorders and administration site conditions | 2
  Vessel puncture site bruise | 2
  Immune system disorders | 1
  Anaphylactic reaction | 1
  Infections and infestations | 1
  Sinusitis | 1
  Musculoskeletal and connective tissue disorders | 1
  Myalgia | 1
  Nervous system disorders | 5
  Dizziness | 2
  Presyncope | 3
  Headache | 1
  Psychiatric disorders | 1
  Anxiety | 1
  Respiratory, thoracic and mediastinal disorders | 2
  Rhinorrhoea | 2
  Oropharyngeal pain | 1
  Vascular disorders | 1
  Hot flush | 1

13. Secondary Outcome: Incidence of Adverse Events of Special Interest (AESI) Through Day 183
Description: Incidence of AESIs Through Day 183
Time Frame: 182 days post vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Participants | 0

14. Secondary Outcome: Incidence of Serious Adverse Events (SAEs) Through Day 183
Description: Incidence of SAEs Through Day 183
Time Frame: 182 days post vaccination
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Time Frame: AEs include solicited AEs collected through Day 8 and unsolicited AEs collected through Day 29. SAEs (reported separately) were collected through Day 183.
Arm/Group | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 17/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PXVX0317 (CHIKV VLP, Alum-adjuvanted) Vaccine (N=25)
Nausea (Gastrointestinal disorders) | 2
Injection site pain (General disorders) | 14
Fatigue (General disorders) | 8
Vessel puncture site bruise (General disorders) | 2
Chills (General disorders) | 1
Pyrexia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Sinusitis (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or release study data after the earlier of (a) the date of publication of a multi-center publication coordinated by Sponsor on the study data, or (b) the date of submission of the study data by Sponsor to regulatory authorities for regulatory approval; provided that PI furnishes Sponsor with a copy of any proposed publication or release at least ninety days in advance of the proposed submission or presentation date for review. PI must acknowledge Sponsor on any publication.

DOCUMENTS (3):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT05065983/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT05065983/SAP_001.pdf
  • Informed Consent Form (2021-12-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT05065983/ICF_002.pdf